CLINICAL TRIAL: NCT01459042
Title: Prevalence of Primary Aldosteronism and Status of Renin-Angiotensin System in Resistant Hypertension:An Observational Study in China
Brief Title: Prevalence of Primary Aldosteronism in Patients With Resistant Hypertension in China
Status: Completed | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Wang Weiqing, Endocrinology Department of Ruijin Hospital affiliated Shanghai Jiao Tong University School of Medicine, Shanghai Jiao Tong University School of Medicine
Other Study IDs: 19830409
Record Dates: First submitted 2011-10-21; First posted 2011-10-25 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Hypertension, Resistant to Conventional Therapy
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood samples,including serum, plasma and whole blood.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- primary aldosteronism
- essential hypertension

SUMMARY:
Recent studies indicate that primary aldosteronism (PA) is a much more common cause of hypertension than had been demonstrated historically. In patients with resistant hypertension, the prevalence of PA from different clinics worldwide is about 10-20%. As has been no such data in China, the investigators are conducting a PA study in different province of China to evaluate the prevalence of PA in patients with resistant hypertension.

ELIGIBILITY:
Inclusion Criteria:

* patients with resistant hypertension
* age 18-65 years

Exclusion Criteria:

* known cause of hypertension
* heart failure
* renal dysfunction
* Stroke, transient ischaemic attack or myocardial infarction in the past 6 months
* cirrhosis
* pregnancy
* undertreatment of glucocorticoid

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with resistant hypertension from different provinces of China
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Weiqing Wang, MD, PhD, Principal Investigator — Endocrinology Department of Ruijin Hospital affiliated Shanghai Jiao Tong University School of Medicine
Locations (1):
- Dep.endocrinology of Shanghai Ruijin Hospital, Shanghai Jiaotong university school of medcine, Shanghai, Shanghai Municipality, China